CLINICAL TRIAL: NCT03031769
Title: Symptoms and Physical Activity in COPD Patients in Europe
Acronym: SPACE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5970R00006
Record Dates: First submitted 2016-12-20; First posted 2017-01-26 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational, multinational, cross sectional study to describe 24-hs symptoms, physical activity and their relationship in stable COPD patients in Europe

DETAILED DESCRIPTION:
The study is a multi-centre, multi country, observational prospective cross sectional study to determine the prevalence and severity of early morning, day and night-time symptoms and physical activity patterns and to evaluate their correlation between each other and with disease severity, adherence to respiratory medications, direct costs and PROs in patients with stable COPD in Europe.

Approximately 2000 patients will be enrolled in convenient sites in several (9-12) selected countries.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 40 years or older.
2. Patient has diagnosis of COPD for 1 year or more.
3. Patient has at least one spirometry with COPD criteria, fixed ratio <0.70 post BD, in previous 12 months
4. Patient is a current smoker or an ex-smoker with a smoking history of ≥ 10 pack- years.
5. Stable patients, as stated in medical records or patient reports during visit, defined as: without exacerbation treatment at study visit neither in the previous 2 months, and without changes in maintenance COPD treatment regimen over the preceding 2 months (avoid first consult patient)
6. Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
7. After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Patient has diagnosis of sleep apnea syndrome or other chronic respiratory disease different from chronic obstructive diseases. (except for non-idiopathic pulmonary fibrosis and ACOS, only if the main diagnosis is COPD)
2. An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to complete questionnaires or participate in this study
3. Patient is participating in an ongoing clinical trial that might, in the investigator's opinion, influence the assessment for SPACE study

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female ambulatory patients aged over 40 years diagnosed with stable COPD according 2013 GOLD criteria
Sampling Method: Non-Probability Sample
Enrollment: 2176 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing symptoms (previous 24 hours) and insufficient physical activity levels (previous month) despite being treated for COPD in real life setting. | Day 1

SECONDARY OUTCOMES:
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and physical activity level (YPAS questionnaire) on day 1 | Day 1
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and adherence to respiratory medication (SRSI for patients and inhalers technique assessed by investigators) on day 1 | Day 1
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and disease classification (By GOLD recommendation) on day 1 | Day 1
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and level of dyspnea level (mMRC) on day 1 | Day 1
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and HRQoL (CAT) on day 1 | Day 1
• Relationship between 24 hours symptoms (Exact, EMSCI & NiSCI questionnaires) and history of exacerbations (By GOLD definition) in last 12 months | Day 1
• Relationship between physical activity levels (YPAS questionnaire) and adherence to respiratory medication (SRSI for patients and inhalers technique assessed by investigators) on day 1 | Day 1
• Relationship between physical activity levels (YPAS questionnaire) and disease classification (By GOLD recommendation) on day 1 | Day 1
• Relationship between physical activity levels (YPAS questionnaire) and level of dyspnea level (mMRC) on day 1 | Day 1
• Relationship between physical activity levels (YPAS questionnaire) and HRQoL (CAT) on day 1 | Day 1
• Relationship between physical activity levels (YPAS questionnaire) and history of exacerbations (By GOLD definition) in last 12 months | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Florin D Mihaltan, MD,PhD, Study Chair — Institute Marius Nasta, Bucharest
Locations (1):
- Research site, Iași, Romania

REFERENCES:
- [Derived] Mihaltan F, Rajnoveanu RM, Arghir OC, Alecu S, Postolache PA. High 24-Hour Respiratory Symptoms and Low Physical Activity in the Stable COPD Romanian Cohort of SPACE Study. Int J Chron Obstruct Pulmon Dis. 2021 Sep 6;16:2533-2544. doi: 10.2147/COPD.S321197. eCollection 2021. PMID 34522093
- [Derived] De Bontridder S, Corhay JL, Haenebalcke C, Fievet F, Etienne I, Vanderhelst E. Correlation of symptoms and physical activity level in chronic obstructive pulmonary disease patients: results from the observational SPACE study. Acta Clin Belg. 2022 Jun;77(3):671-678. doi: 10.1080/17843286.2021.1950419. Epub 2021 Jul 12. PMID 34252000
- [Derived] Mihaltan F, Adir Y, Antczak A, Porpodis K, Radulovic V, Pires N, de Vries GJ, Horner A, De Bontridder S, Chen Y, Shavit A, Alecu S, Adamek L. Importance of the relationship between symptoms and self-reported physical activity level in stable COPD based on the results from the SPACE study. Respir Res. 2019 May 14;20(1):89. doi: 10.1186/s12931-019-1053-7. PMID 31088560